CLINICAL TRIAL: NCT04753086
Title: LCCC 2052: Patient Related Outcomes for Gynecologic Radiation Oncology (PRO-GRO)
Brief Title: Patient Related Outcomes for Gynecologic Radiation Oncology
Acronym: PRO-GRO
Status: Active, not recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 2052
Record Dates: First submitted 2021-02-03; First posted 2021-02-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologic Cancer Pts: Gynecologic cancer patients being treated with radiation at UNC.

SUMMARY:
The goal of this study is to see if it is feasible to use electronic questionnaires to measure patient related outcomes before, during, and after radiation for gynecologic cancer in a high-volume radiation oncology clinic.

DETAILED DESCRIPTION:
Other studies have found benefits from using patient related outcome measurements (PROM) in clinical settings, and a paper PROM is part of standard of care treatment for prostate cancer patients at the University of North Carolina clinic. However, PROM are not routinely collected for gynecological cancer patients at UNC, and fewer studies have specifically focused on PROM for gynecological cancer patients receiving radiation. The primary objective of this study is to determine the feasibility of PRO monitoring of gynecologic symptoms before, during (at weekly intervals), and after radiation (external beam radiotherapy and brachytherapy) for gynecologic cancer patients at a high volume center.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Informed consent reviewed and signed
* Gynecologic cancer being treated by radiation at UNC
* Able and willing to complete web-based symptom survey

Exclusion Criteria:

* Inability to read and speak English
* Current incarceration
* Pregnancy
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rending of informed consent (with the caveat that if they initially are hospitalized with delirium which is subsequently resolved, they can then be consented for participation at a later time)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecologic cancer receiving radiation treatment at the University of North Carolina
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Rate of survey completion at acute timepoints | First week of radiation to 6 weeks after completing radiation
  Percentage of patients who complete at least 75% of the questionnaires given after the baseline and up to and including the 6-week post-treatment survey

SECONDARY OUTCOMES:
Rate of survey completion at late timepoints | 6 months post-treatment to 2 years post-treatment
  Percentage of patients who complete at least 75% of the questionnaires given after and including the 6-month post-treatment survey and up to and including the 2-year post-treatment survey
Late, persistent, substantial, treatment-related symptoms (LAPERS) | 6 months post-treatment to 2 years post-treatment
  LAPERS will only be calculated for patients who have baseline symptoms (actual baseline or 3 months post-treatment, whichever is lower), one early follow up assessment (1, 2, or 6 week post-treatment), and at least 3 late follow ups (6 months post-treatment or later). If a patient's symptom worsened to "quite a bit" or "very much" in at least half of the late follow-ups, this will be considered LAPERS. Thus LAPERS is a binary score that will be assessed for each symptom in each patient.
Incidence of acute symptoms for all patients | First week of radiation to 6 weeks after completing radiation
  We will calculate incidence of each symptom, for all patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of acute symptoms for all patients | First week of radiation to 6 weeks after completing radiation
  We will calculate prevalence of each symptom, for all patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of acute symptoms for all patients | First week of radiation to 6 weeks after completing radiation
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of late symptoms for all patients | 6 months post-treatment to 2 years post-treatment
  We will calculate incidence of each symptom, for all patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of late symptoms for all patients | 6 months post-treatment to 2 years post-treatment
  We will calculate prevalence of each symptom, for all patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of late symptoms for all patients | 6 months post-treatment to 2 years post-treatment
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of acute symptoms for cervical cancer patients | First week of radiation to 6 weeks after completing radiation
  We will calculate incidence of each symptom for cervical cancer patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of acute symptoms for cervical cancer patients | First week of radiation to 6 weeks after completing radiation
  We will calculate prevalence of each symptom for cervical cancer patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of acute symptoms for cervical cancer patients | First week of radiation to 6 weeks after completing radiation
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of late symptoms for cervical cancer patients | 6 months post-treatment to 2 years post-treatment
  We will calculate incidence of each symptom for cervical cancer patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of late symptoms for cervical cancer patients | 6 months post-treatment to 2 years post-treatment
  We will calculate prevalence of each symptom for cervical cancer patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of late symptoms for cervical cancer patients | 6 months post-treatment to 2 years post-treatment
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of acute symptoms for endometrial cancer patients | First week of radiation to 6 weeks after completing radiation
  We will calculate incidence of each symptom for endometrial cancer patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of acute symptoms for endometrial cancer patients | First week of radiation to 6 weeks after completing radiation
  We will calculate prevalence of each symptom for endometrial cancer patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of acute symptoms for endometrial cancer patients | First week of radiation to 6 weeks after completing radiation
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of late symptoms for endometrial cancer patients | 6 months post-treatment to 2 years post-treatment
  We will calculate incidence of each symptom for endometrial cancer patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of late symptoms for endometrial cancer patients | 6 months post-treatment to 2 years post-treatment
  We will calculate prevalence of each symptom for endometrial cancer patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of late symptoms for endometrial cancer patients | 6 months post-treatment to 2 years post-treatment
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of acute symptoms for vulvar cancer patients | First week of radiation to 6 weeks after completing radiation
  We will calculate incidence of each symptom for vulvar cancer patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of acute symptoms for vulvar cancer patients | First week of radiation to 6 weeks after completing radiation
  We will calculate prevalence of each symptom for vulvar cancer patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of acute symptoms for vulvar cancer patients | First week of radiation to 6 weeks after completing radiation
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.
Incidence of late symptoms for vulvar cancer patients | 6 months post-treatment to 2 years post-treatment
  We will calculate incidence of each symptom for vulvar cancer patients. Incidence is defined as the number of patients who have a symptom in any follow up.
Prevalence of late symptoms for vulvar cancer patients | 6 months post-treatment to 2 years post-treatment
  We will calculate prevalence of each symptom for vulvar cancer patients. Prevalence is the number of patients with a given symptom at a set time point.
Time course of late symptoms for vulvar cancer patients | 6 months post-treatment to 2 years post-treatment
  We will evaluate the time course by creating a graphical representation of each symptom severity at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Weiner, M.D., Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States